CLINICAL TRIAL: NCT04354870
Title: Off Label Study to Evaluate the Efficacy of HCQ for Pre-exposure Prophylaxis (PrEP) to Prevent Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection Among Health Care Workers (HCWs) Who Are at High Risk of Occupational Exposure to SARS-CoV-2
Brief Title: COVID-19 PrEP HCW HCQ Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: s20-00390
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Results first posted 2021-10-06 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Total number of participant: 350 (Group A and B)
  * Group A: projected 300 (HCW choose to be provided HCQ)
  * Group B: projected 50 (HCW choose not to be provided HCQ)
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HCQ Group (Experimental): Approximately 300 Health Care Workers (HCW) who choose to be provided HCQ
  Interventions: Drug: Hydroxychloroquine (HCQ)
- Control Group (No Intervention): approximately 50 HCW who choose not to be provided HCQ

INTERVENTIONS:
Drug: Hydroxychloroquine (HCQ) — Loading dose: 600 mg, oral, 1 day Maintenance dose: 200 mg, oral, daily, for 90 days
  Arms: HCQ Group

SUMMARY:
Off label study to evaluate the efficacy of HCQ for pre-exposure prophylaxis (PrEP) to prevent severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection. 350 participants will be assigned to the group that takes HCQ or the group that opts to not take the study medication. Participants will be NYULH HCW at high risk for occupational exposure to SARS-CoV-2. Study timepoints will include screening/enrollment, 30 day, 60 day, and 90 day visits. Questionnaires, and DBS will be collected in all timepoints.

DETAILED DESCRIPTION:
Hydroxychloroquine (HCQ) is licensed for the chemoprophylaxis and treatment of malaria and as a disease modifying antirheumatic drug. It has a long history of being safe and well tolerated at typical doses. HCQ has antiviral activity in vitro against coronaviruses, and specifically Covid-19. This study is designed to evaluate the efficacy of hydroxychloroquine (HCQ) for pre exposure prophylaxis (PrEP) to prevent severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection among health care workers at high risk of occupational exposure to SARS-CoV-2 compared to the eligible cohort that declines treatment.

ELIGIBILITY:
Inclusion Criteria for Group A and B

* Men or women ages ≥18 years NYULH health care worker who meets one of the following criteria

  1. Involved in an aerosol generating procedure (nasopharyngeal specimen collection, tracheal intubation, nebulizer treatment, open airway suctioning, collection of sputum, tracheostomy, bronchoscopy, CPR) on a confirmed COVID-19 patient while wearing PPE
  2. Direct bedside care of confirmed COVID-19 patient while wearing PPE for 3 or more shifts in a 7 day period
  3. Direct care of PUIs in the ED or other inpatient unit while wearing PPE for 3 or more shifts in a 7 day period
* Willing and able to provide informed consent

Exclusion Criteria for Group A only :

* Known hypersensitivity to hydroxychloroquine or chloroquine
* Known diagnosis of COVID-19
* Concomitant use of

  1. amiodarone
  2. digoxin
  3. flecainide
  4. procainamide
  5. propafenone
* History of Torsades de pontes
* History of retinal disease
* Known chronic kidney disease ≥ stage 4
* Congenital prolonged QTc interval syndrome (Jervell and Lange-Nielsen syndrome, Romano-Ward syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Michael Belmont, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Study internal to NYU at this time

REFERENCES:
- [Result] Raabe VN, Fleming A, Samanovic MI, Lai L, Belli HM, et al. (2022) Hydroxychloroquine Pre-Exposure Prophylaxis to Prevent SARS-CoV-2 Among Health Care Workers at High Risk For SARS-CoV-2 Exposure: A Nonrandomized Controlled Trial. Infect Dis Diag Treat 6: 201.
- See also: DOI: https://doi.org/10.29011/2577-1515.100201. — https://www.gavinpublishers.com/article/view/hydroxychloroquine-pre-exposure-prophylaxis-to-prevent-sars-cov-2-among-health-care-workers-at-high-risk-for-sars-cov-2-exposure-a-nonrandomized-controlled-trial

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HCQ Group | Control Group
Started | 83 | 47
Completed | 35 | 14
Not Completed | 48 | 33
Not completed — Lost to Follow-up | 32 | 12
Not completed — Withdrawal by Subject | 10 | 16
Not completed — Did not complete all study visits | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HCQ Group | Control Group | Total
Number analyzed (Participants) | 35 | 14 | 49
Age, Continuous [Mean (Full Range); unit: years] | 43.6 [27 to 65] | 43.7 [25 to 63] | 43.7 [25 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 9 | 28
  Male | 16 | 5 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 33 | 14 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 27 | 9 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Number of Participants With Seroconversion to SARS-CoV-2 at 1 Month
Description: Antibody titers will be measured to determine seroconversion, a binomial endpoint defined by a four-fold increase in antibody titers compared to baseline.
Time Frame: Baseline to 1 month post-baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HCQ Group | Control Group
Number analyzed (Participants) | 56 | 24
Participants | 4 | 2

2. Primary Outcome: Number of Participants With Symptomatic vs. Asymptomatic Seroconversion
Description: To characterize whether high-risk HCW who seroconvert to SARS-CoV-2 have asymptomatic infection or report symptoms of COVID-19 in the 4 weeks preceding seroconversion (assessed by symptom questionnaire).
Time Frame: 4 Weeks Prior to Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | HCQ Group | Control Group
Number analyzed (Participants) | 56 | 24
Participants
  Symptomatic Seroconversion | 1 | 2
  Asymptomatic Seroconversion | 3 | 0

3. Secondary Outcome: Number of Participants With of AEs or SAEs Possibly, Probably, or Definitely Related to HCQ Upon Study Termination Time
Description: To assess the tolerability of hydroxychloroquine SARS-CoV-2 PrEP in this population
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | HCQ Group | Control Group
Number analyzed (Participants) | 83 | 47
Participants
  with AEs Related to HCQ | 8 | 0
  with SAEs Related to HCQs | 0 | 0

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | HCQ Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/47
Other Adverse Events (participants affected / at risk) | 8/83 | 0/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HCQ Group (N=83) | Control Group (N=47)
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Itching (Skin and subcutaneous tissue disorders) | 1 | 0
Hair Loss (General disorders) | 1 | 0
Appetite Loss (General disorders) | 1 | 0
Gastrointestinal Discomfort (Gastrointestinal disorders) | 1 | 0
Gastroesophageal Reflux (Gastrointestinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT04354870/Prot_SAP_000.pdf